CLINICAL TRIAL: NCT05498103
Title: Use of Methazolamide to Lower Intraocular Pressure
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0721
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Glaucoma, Open-Angle
Keywords: Glaucoma; Methazolamide; Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Methazolamide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methazolamide 25 mg (Active Comparator): Once a day [q.d] in the morning for 1 week, Twice a day [b.i.d.] in the morning and evening for 1 week
  Interventions: Drug: Methazolamide 25 MG
- Methazolamide 50 mg (Active Comparator): Once a day [q.d] in the morning for 1 week, Twice a day [b.i.d.] in the morning and evening for 1 week
  Interventions: Drug: Methazolamide 50 MG

INTERVENTIONS:
Drug: Methazolamide 25 MG — 25 mg tablets
  Arms: Methazolamide 25 mg
Drug: Methazolamide 50 MG — 50 mg tablets
  Arms: Methazolamide 50 mg

SUMMARY:
The purpose of this study is to evaluate the effect of methazolamide, 25 mg or 50 mg tablets once a day for a week than twice a day for a week, on lowering intraocular pressure and the safety of methazolamide.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 50 and 90 years old
* Current diagnosis of open angle glaucoma (OAG) in both eyes
* Ability to read and write in English

Exclusion Criteria:

* Glaucoma other than OAG
* Severe or end-stage glaucoma (cup to disc ratio >0.8 or Mean Deviation on Visual Field worse than -12)
* Pregnant or breast-feeding women

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percent IOP change at each follow-up Visit | Day 1 (Pre-dosing, then 4- and 8- hours post dosing), Day 7 (Pre-dosing, then 4- and 8- hours post dosing), Day 14 (Pre-dosing, then 4- and 8- hours post dosing)
  IOP measure is measured using Goldmann Tonometry. IOP is measured in mmHg with a normal range from 12 mmHg to 22 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y. Kahook, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Sue Anschutz-Rodgers Eye Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No